CLINICAL TRIAL: NCT06771440
Title: Impact Assessment of a Clinical Decision Support Tool for Non-invasive Antibiotic Allergy Label Delabeling and Refinement
Brief Title: Support Tool for Antibiotic Allergy deLabeling
Acronym: STAAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Noorderhart Pelt (Other); AZ Herentals (Unknown); Heilig Hartziekenhuis, Mol (Unknown); AZ Turnhout (Other); Sint-Jozefskliniek Izegem (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: S68439
Record Dates: First submitted 2024-12-20; First posted 2025-01-13 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2024-12

CONDITIONS: Antibiotic Allergy
Keywords: Penicillin allergy; Delabeling; beta-lactam; electronic health records; clinical decision support; Antibiotic allergy; drug allergy
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Multi-centre open label cross-over cluster-randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AAL fact-check (Experimental): Semi-automated EPR search for re-exposure
  Interventions: Other: EPR search
- Standard of care (no AAL fact-check) (No Intervention)

INTERVENTIONS:
Other: EPR search — A stored query in the EPR, that checks for re-exposure to the culprit antibiotic or class-member, from the date of AAL registration to the date of patient inclusion
  Other Names: AAL-fact-check tool
  Arms: AAL fact-check

SUMMARY:
Antibiotic allergy labels (AAL) are reported in 7% of inpatient's charts, especially for beta-lactams (86% of AAL, i.e., prevalence of 6%). They are associated with increased length of hospital stay, and use of second-line and broad-spectrum antibiotics. Allergy workups are able to invalidate the majority of these AAL but are time-consuming and require invasive skin and provocation testing. The investigators recently evaluated, for the first time in Europa, a strictly non-invasive delabeling protocol using a questionnaire, medical file search and contact with primary care health care workers in 200 adult internal medicine inpatients with a beta-lactam AAL. Up to half of the AAL could be removed or refined, demonstrating the potential of this strategy. In this project, they aim to assess the impact of using the non-invasive 'AAL-fact-check' tool in a multicenter study, on antibiotic selection, and clinical, antimicrobial, and economic endpoints, as compared with the standard of care (i.e., no AAL-fact-check tool).

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patients
2. AAL for one or more beta-lactams

Exclusion Criteria:

1. Age younger than 18
2. Previous enrolment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
First line antibiotic use: yes (1)/no (0) | Until 100 days after discharge
  First line and/or narrow-spectrum beta-lactam antibiotic use (depending on the index indication, and following the guidelines of the Belgian Antibiotic Policy Coordination Commission BAPCOC), as a binary outcome.

SECONDARY OUTCOMES:
Antibiotic allergy label removed: yes (1)/no (0) | Until 100 days after discharge
Antibiotic allergy label refined: yes (1)/no (0) | Until 100 days after discharge
Beta-lactam antibiotic tolerance: yes (1)/no (0) | Until 100 days after discharge
Need to switch antibiotics: yes (1)/no (0) | Until 100 days after discharge
Days until clinical recovery (days) | Until 14 days after discharge
In-hospital mortality: yes (1)/no (0) | Until 14 days after discharge of discharge/death
3 months post-hospitalization mortality: yes (1)/ no (0) | Until 14 days after discharge
Length of hospital stay (days) | Until 14 days after discharge
  Calculated as (date of discharge) - (date of admission) + 1
Admission to ICU: yes (1)/no (0) | Until 14 days after discharge
Readmission within 3 months after discharge: yes (1)/no (0) | Until 100 days after discharge
Colonization with MRSA: yes (1)/no (0) | Until 100 days after discharge
Infection with MRSA: yes (1)/no (0) | Until 100 days after discharge
Colonization with VRE: yes (1)/no (0) | Until 100 days after discharge
Infection with VRE: yes (1)/no (0) | Until 100 days after discharge
Colonization with C.Diff: yes (1)/no (0) | Until 100 days after discharge
Infection with C.Diff: yes (1)/no (0) | Until 100 days after discharge
Cost of antibiotic treatment (euro) | Until 14 days after discharge
Cost of hospitalization (euro) | Until 14 days after discharge
Time needed to perform the AAL fact-check (minutes) | Until 14 days after discharge
  AAL fact-check procedure will be timed by the investigator
Cost of human resources needed for AAL-fact-check (euro) | Until 14 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Rik Schrijvers, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium